CLINICAL TRIAL: NCT01454609
Title: Safety and Efficacy of Bilateral Superficial Cervical Plexus Block in Thyroidectomy - a Double Blind Randomized Controlled Trial
Brief Title: Safety and Efficacy of Bilateral Superficial Cervical Plexus Block in Thyroidectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Principal Investigator, Karthikeyan V S, Senior Resident, Urology, Jawaharlal Institute of Postgraduate Medical Education & Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 100745483-1910201028464726
Record Dates: First submitted 2011-10-08; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Pain; Postoperative
Keywords: cervical plexus block; thyroidectomy; postoperative analgesia
MeSH Terms: conditions — Pain | interventions — Saline Solution; Sodium Chloride; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saline (Placebo Comparator): 0.9% normal saline
  Interventions: Drug: 0.9% Normal saline
- Bupivacaine (Experimental): 0.25% bupivacaine
  Interventions: Drug: Bupivacaine
- Bupivacaine with clonidine (Experimental): 0.25% bupivacaine with 1 microgram/kg of clonidine
  Interventions: Device: Bupivacaine with clonidine (combination)

INTERVENTIONS:
Drug: 0.9% Normal saline — Saline
  Other Names: Saline
  Arms: Saline
Drug: Bupivacaine — Bupivacaine - amide local anesthetic, maximum recommended dose is 2 mg/kg duration 2 - 4 hours of sensory anesthesia up to 24 hours
  Other Names: Marcaine; Sensoricaine
  Arms: Bupivacaine
Device: Bupivacaine with clonidine (combination) — Bupivacaine - amide local anesthetic, maximum recommended dose is 2 mg/kg duration 2 - 4 hours of sensory anesthesia up to 24 hours
  Clonidine - 0.5 - 1 microgram/ kg
  Other Names: Marcaine (for bupivacaine); Sensoricaine (for bupivacaine)
  Arms: Bupivacaine with clonidine

SUMMARY:
With thyroid surgery being performed as an ambulatory procedure, most recent studies concerning post thyroidectomy analgesia are focused on regional techniques such as bilateral superficial cervical plexus block (BSCPB) and bilateral combined superficial and deep cervical plexus block. But, data regarding the efficacy of BSCPB are controversial. Hence the investigators compared the efficacy of BSCPB with 0.25% bupivacaine with or without clonidine in thyroidectomy, as preemptive analgesia.

The hypothesis was bupivacaine with the addition of clonidine would help in reducing postoperative pain and thereby reduce the need for postoperative analgesia.

DETAILED DESCRIPTION:
To find out if addition of BSCPB to general anesthesia with bupivacaine with or without clonidine prolongs the time needed for postoperative analgesic and facilitate to perform thyroidectomy as a day care procedure and to see if clonidine reduces postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Consenting consecutive euthyroid patients undergoing elective thyroidectomy under general anesthesia, of either genders and more than 18 years of age, belonging to the ASA class I and II.

Exclusion Criteria:

* Patients unable to understand visual analog pain score (VAS) or unable to use patient controlled analgesia (PCA).
* Patients with malignancy requiring block dissection or with substernal goiters - Contraindications to superficial cervical plexus block like allergy to local anesthetics, bleeding diatheses and local infection or sepsis.
* Contraindications to morphine like bronchial asthma and hypothyroidism.
* Sensitivity to the anesthetic agent used or intolerance to the medications used in the study.
* Patients who received steroids or opioids or other analgesics recently.
* Patients with history of stridor.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Intraoperative fentanyl requirement and the total morphine requirements in the 24-hour postoperative period | Intraoperative to 24 hours postoperative

SECONDARY OUTCOMES:
Visual analog pain scores at specific time intervals | 24 hours postoperative
Postoperative nausea and vomiting (PONV)and anti emetic requirements | 24 hours postoperative
Side effects of the block, morphine and clonidine | 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Sarath Chandra Sistla, MS(Surgery), Study Chair — Professor, Dept. of Surgery, JIPMER
Locations (1):
- Jawaharlal Institute of Postgraduate Medical Education and Research, Puducherry, Puducherry, India